CLINICAL TRIAL: NCT05009719
Title: Study of the Efficacy and Safety of Risk-adapted Donor Lymphocyte Infusions for the Prophylaxis and Prevention of Relapses After Allogeneic Hematopoietic Stem Cell Transplantation in Children and Adolescent With Hematologic Malignancy
Brief Title: Risk-adapted Donor Lymphocyte Infusion After Allo-HSCT in Children With Hematologic Malignancy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science RM Gorbacheva Institute, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: hsct/dli
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hematologic Malignancy
Keywords: allo-HSCT; children; Donor LymphocyteI Infusion
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: The patients in this study will be divided into 2 groups: prophylactic and preventive depending on indications. Patients without signs of disease with high risk of relapse will be included into prophylactic group. Patients with persistence minimal residual disease or cytogenetic relapse will be included into preventive group. Also, patients will move from the first group to second group, if the clinical status changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic (Experimental): The patients with high risk of relapse of disease and full donor chimerism after allo-HSCT without signs of the disease will be include in this group.
  Interventions: Biological: Prophylactic Donor lymphocytes infusions
- Preventive (Experimental): The patients with persisted minimal residual disease or cytogenetic relapse after allo-HSCT will be include in this group.
  Interventions: Biological: Preventive Donor lymphocytes infusions

INTERVENTIONS:
Biological: Prophylactic Donor lymphocytes infusions — Donor lymphocytes is taken by apheresis or dose of blood from allogeneic donor. After apheresis lymphocytes arel freezed for next using. DLI is transfused to patients IV using central venous access.
  Donor lymphocytes infusion start from D+60 - D+100 and continue with escalating doses every 1.5-3 months during first year after HSCT up to appearance of GVHD or signs of disease. First dose is 1*10*6 CD3+/kg. Subsequent doses increases by 0.5 log for haploidentical and unrelated donor and 1 log for sibling donor up to 1*10*8 CD3+/kg.
  Arms: Prophylactic
Biological: Preventive Donor lymphocytes infusions — Donor lymphocytes is taken by apheresis or dose of blood from allogeneic donor. After apheresis lymphocytes freeze for next using. DLI are transfused to patients IV using central venous access.
  Donor lymphocytes infusion continue with escalating doses every 1.5-3 months up to achieving MRD negative status or appearance of GVHD or signs of active disease.
  First dose is 1*10*6 CD3+/kg for patients without previous GVHD and 1*10*5 CD3+/kg for patients with previous GVHD. Subsequent doses increases by 0.5 log for haploidentical and unrelated donor and 1 log for sibling donor up to 1*10*8 CD3+/kg.
  Arms: Preventive

SUMMARY:
Allo-hsct is potentially curative method of treatment for children and adolescent with hematologic malignancy. However, relapses of disease after allo-hsct occur up to 50% of patients and constitute the main cause of mortality after HSCT. Donor lymphocytes infusion (DLI) is a form of immunotherapy based on developement of reaction "graft versus from leukemia". This study evaluates the safety and efficacy of risk-adapted srtategy of DLI for prophylaxis and prevention posttransplant relapses in children and adolescent with hematologic malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 months - 18 years old
* Diagnosis: acute lymphoblastic leukemia, acute myeloid leukemia, juvenile myelomonocytic leukemia, myelodysplastic syndrome, chronic myeloid leukemia
* Signed by legal representatives informed consent
* High risk disease ( for ALL - initial hyperleukocytosis> 50x109 / L, T-cell ALL, hypodiploid karyotype, complex karyotype, MLL gene rearrangement, SIL-TAL deletion, primary resistent of the disease, early/very earle relapse, infant ALL; for AML patients - rearrangement of the MLL gene (except for t (1; 11) and t (9; 11) with M5 morphology), inv (3), t (3; 3), complex karyotype anomalies, t (8; 21 ) with trisomy 4, t (16; 21), monosomy 7, monosomy 5, M7 without t (1; 22), FLT3+, M6, t (7; 12), AML with multilineage dysplasia, p53 gene mutations, NUP98 translocations, primary resistent of the disease, early/very earle relapse infant AML, secondary AML; all juvenile myelomonocytic leukemia and myelodysplastic syndrome; allo-HSCT at 3 or more remission; persistence MRD before alloHSCT; allo-HSCT out of remission; persistence MRD after alloHSCT; cytogenetic relapse after alloHSCT )
* Donor chimerism=>95%
* No poor graft function (haemoglobin concentration < 100 g/L; neutrophils < 1.0 × 10E + 9/L; and platelets < 30 × 10E + 9/L on day ≥ 30 post transplant with complete donor chimerism and no graft-versus-host disease or relapse )
* ECOG 0-2 status
* Karnofsky/Lansky status >30%

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Severe organ failure: creatinine more than 2 norms; ALT, AST more than 5 norms; bilirubin more than 1.5 norms
* Ejection fraction less than 50%
* Requirement for vasopressor support at the time of enrollment
* Somatic or psychiatric disorder making the patient unable to sign an informed consent
* Acute GVHD grade 3-4 in patient medical history
* Severe chronic GVHD in patient medical history

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Relapse - free survival | 24 months
  Estimate time to morphological relapse by Kaplan Mayer

SECONDARY OUTCOMES:
Overall survival analysis | 24 months
  Estimate time to death by Kaplan Mayer
Relapse rate analysis | 24 months
  Cumulative incidence of patients with relapse by Gray's test
Non-relapse mortality analysis | 24 months
  Cumulative incidence of patients with mortality without hematological relapse of malignancy
Incidence of acute GVHD grade II-IV | 125 days
  Cumulative incidence of patients with acute GVHD II-IV grade by Gray's test
Incidence of moderate and severe chronic GVHD | 24 months
  Cumulative incidence of patients with moderate and severe chronic GVHD according to NIH 2015 criteria by Gray's test
Incidence of achievement MRD negative status | 24 months
  Cumulative incidence of patients with MRD positive status, who had responds to therapy Gray's test
Relapse - free survival | 24 months
  Estimate time to appearing of MRD or morphological relapse by Kaplan Mayer
Graft - versus -host-disease free/relapse free survival | 24 months
  Estimate time to date of III-IV acute GVHD (aGVHD), chronic GVHD (cGVHD) requiring systemic immunosuppressive treatment, disease relapse or death from any other cause by Kaplan Mayer

CONTACTS AND LOCATIONS:
Locations (1):
- RM Gorbacheva Research Institute, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No